CLINICAL TRIAL: NCT06059768
Title: Urdu Translation and Psychometric Analysis of Lawton Instrumental Activities of Daily Living Scale.
Brief Title: Urdu Translation and Psychometric Analysis of Lawton IADLS.
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: RiphahIU Rida Maryaum
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Cognitive Dysfunction
Keywords: Cognitive Dysfunction, Geriatrics, Psychometric, Validity
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Functional capacity and independent living skills are most crucial and important aspects to measure in older adults. Lawton IADL is an 8-item scale used to assess independent living skills. Lawton IADLS was originally developed in English. It has been translated and validated in several languages and showed excellent reliability and responsiveness. In our study Lawton IADL scale will be translated in Urdu and its psychometric analysis will be performed.The study design will be descriptive translation study. Study will be conducted in Rahimoon Welfare Foundation old age home of Lahore. Inclusion criteria will be patients of age between 65-75 years with both genders scoring 24 or more on MMSE and those who will be fluent in Urdu language. Those patients will be excluded who will have neurological problems affecting their IADLS, Cognitive/communication dysfunction or Patients with musculoskeletal impairments affecting IADLs. Participants will be asked to perform Lawton IADLs on the instruction and on completion performance will be scored. Study will be completed in two phases. Phase I will consist of Translation of original version (English) into Urdu version and pilot-testing of translated version. In phase II psychometric analysis will be performed. Data will be analyzed using SPSS version 21.

DETAILED DESCRIPTION:
Aging is a constant, natural and inevitable process in living creatures' lives, characterized by bio psychosocial and cultural changes that are affected by intrinsic factors such as genetics and by extrinsic factors such as acquired experiences and the environment (World Health Organization [WHO], 2010).

Geriatrics refers to medical care for older adults, there is no set age to define older age, but age greater than 65 is mostly used. The elderly, or those older than 65 years, currently represent 12.5 percent of the U.S. population.With increasing life spans across the world, Pakistan is also experiencing a rise in its elderly population.According to 1998 Census report, in Pakistan the population of over-60 years increased to 7.34 million .Functional capacity is a complex concept that includes basic activities of daily living (BADL), instrumental activities of daily living (IADL),and advanced activities.BADL demonstrate the effectiveness of rehabilitation, and determine a person's ability to perform activities of daily living.The BADL may decline due to age, a specific disease, or a variety of factors such as decreased muscle strength, loss of vision, and postural changes Functional decline in older people is nearly 12% in those more than 75 years of age. According to (ECHP) people over 65 in the European Community, it is observed that 21% of the population is severely deteriorated to carry out activities of daily living, and this figure rises up to 29% for people over 75 years old. France would be the European country with most dependence in the ADL (28% of people over 65). The estimate of prevalence of physical disability in older adults of Punjab Pakistan varied from 13.9% to 36.6%.The assessment of functional status is critical when caring for older adults. A functional assessment can also guide the clinician to focus on the person's baseline capabilities, facilitating early recognition of changes that may signify a need either for additional resources or for a medical work-up. number of questionnaires are available to assess IADL, however, no gold standard exists . One of the most widely used is the Lawton Instrumental Activities of Daily Living Scale developed in 1969 by Lawton and Broady. Lawton IADL is an 8-item scale used to assess independent living skills. It is most useful for identifying how a person is functioning at a present time and to identify improvement or deterioration over time.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65-75 years
* Both gender Male and Female
* Sufficient cognitive ability to understand and read the questionnaire with
* MMSE 24 or more.
* Fluent in Urdu Language

Exclusion Criteria:

* Patients with neurological problems affecting their IADLs
* Cognitive/communication impairment.
* Patients with musculoskeletal impairments affecting IADLs

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Subjects with above mentioned inclusion criteria will be taken. Written informed consent will be obtained from all participants. After obtaining demographic data all the participants will be asked to perform Lawton IADLs on the instruction and on completion performance will be scored.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Lawton IADL | 8 months
  It is an 8-item scale used to assess independent living skills. It is most useful for identifying how a person is functioning at a present time and to identify improvement or deterioration over time. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent).Total administration time is 10-15 minutes
Functional Activities Questionnaire | 8 months
  It is a 10 item scale used to measures instrumental activities of daily living scale in older adults. This instrument also measures functional changes over the period of time. Participants respond to 10-items to daily tasks needed when living independently. A scale ranging from independence (0) to dependence (3) is used for responses. Approximately 10 minutes are required for test completion.

SECONDARY OUTCOMES:
Reliability of translated version of Lawton IADLS | 8 months
  The reliability of translated version of Lawton IADLS will be determined by assessing test-retest reliability across repeated measures and internal consistency through crohnbach alpha.
Validity of translated version of Lawton IADLS | 8 months
  Validity is how accurate the results are. Validity of translated version of Lawton IADLS will be determined by assessing face validity by percentage agreement, content validity by CVI and criterion/concurrent validity by Pearson's correlation between Lawton IADLS and FAQ (functional activity questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Rida Maryaum, MSPT-NM, Principal Investigator — Riphah International University
Locations (1):
- Tehreem Mukhtar, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No